CLINICAL TRIAL: NCT02417857
Title: Quality-of-life, Body Image and Cosmesis After Single Incision Laparoscopic Cholecystectomy (SILC) Versus Conventional Laparoscopic Cholecystectomy (CLC)
Brief Title: Comparison of Single İncision Laparoscopic Cholecystectomy Versus Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Mevki Military Hospital (Other)
Responsible Party: Principal Investigator, MD. Mehmet SAYDAM (General Surgeon), General Surgeon (M.D.), Ankara Mevki Military Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMMA-LEC-1648.4-70
Record Dates: First submitted 2015-04-08; First posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Laparoscopic Surgical Procedures
Keywords: Single İncision Laparoscopic Surgery; Conventional Laparoscopic Surgery
MeSH Terms: interventions — Cholecystectomy, Laparoscopic; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Cholecystectomy (SILC) (Experimental): Group 1: Single Incision Laparoscopic Cholecystectomy (Intervention)
  Interventions: Procedure: Laparoscopic Cholecystectomy (Single Incision)
- Laparoscopic Cholecystectomy (CLC) (Experimental): Group 2: Conventional Laparoscopic Cholecystectomy (Intervention)
  Interventions: Procedure: Laparoscopic Cholecystectomy (Conventional)

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy (Single Incision) — We performed Single Incision Laparoscopic Cholecystectomy (SILC) operation to the group-1
  Arms: Laparoscopic Cholecystectomy (SILC)
Procedure: Laparoscopic Cholecystectomy (Conventional) — We performed Conventional Laparoscopic Cholecystectomy (CLC) to group-2
  Arms: Laparoscopic Cholecystectomy (CLC)

SUMMARY:
The aim of this study is to compare outcomes of quality-of-life measures and evaluate the body image and cosmesis between Single Incision Laparoscopic Cholecystectomy (SILC) and Conventional Laparoscopic Cholecystectomy (CLC).Twenty eight patients underwent SILC and 30 underwent LC.Fifty-eight patients were included the study and divided into two groups. The results of the questionnaires were statistically compared.

DETAILED DESCRIPTION:
Recently, single incision laparoscopic cholecystectomy (SILC) is one of the minimally invasive technique, developed to reduce the need of multiple ports and has become popular among the surgeons. This study was conducted with fifty eight patients between January 2011 and March 2013 in Turkey. Fifty-eight patients were included the study and divided into two groups. Quality-of-life measures was evaluated by the EuroQol EQ-5D questionnaire.Cosmesis and body image were evaluated with the Body Image Questionnaire. All statistical analyses were performed by IBM Statistics 21.0 and MS-Excel 2007. A value of p<0.05 was accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* The patients who were scheduled for elective cholecystectomy were included in the study

Exclusion Criteria:

* pregnancy
* acute cholecystitis
* ASA 3-4 (American Society of Anesthesiologists)
* history of bile duct stone migration
* biller pancreatitis
* upper laparatomy
* any ventral hernia repair
* chronic systemic disease or
* with allergic attitude to any agent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Quality of life measure | We had performed the questionnaire at postoperative 6 th month

SECONDARY OUTCOMES:
Body Image Questionnaire measure | We had performed the questionnaire at postoperative 6 th month

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin SINAN, Prof. M.D., Study Director — VAN MILITARY HOSPITAL, GENERAL SURGERY DEPARTMENT, VAN, TURKEY

REFERENCES:
- [Result] Abd Ellatif ME, Askar WA, Abbas AE, Noaman N, Negm A, El-Morsy G, El Nakeeb A, Magdy A, Amin M. Quality-of-life measures after single-access versus conventional laparoscopic cholecystectomy: a prospective randomized study. Surg Endosc. 2013 Jun;27(6):1896-906. doi: 10.1007/s00464-012-2625-5. Epub 2012 Dec 27. PMID 23269370